CLINICAL TRIAL: NCT04612985
Title: Evaluation of the Safety, Effectiveness and Usability of the XACT Robotic System for Image Guided Percutaneous Lung Procedures
Brief Title: Evaluation of the XACT Robotic System for Image-guided Percutaneous Lung Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The IDE wasn't approved
Sponsor: Xact Robotics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-002-00
Record Dates: First submitted 2018-02-14; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: CT-guided Minimally Invasive Procedures e.g. Biopsies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Procedures with XACT Robotic System (Experimental): Device: XACT Robotic System The XACT device is a real-time, CT image guided, 3-dimensional robotic system. The XACT device is intended for use as an image guided positioning and steering system for insertion of clinical tools, such as biopsy needles, ablation needles, etc., during minimally invasive percutaneous lung procedures. The system is defined to guide (i.e., position and steer) the tool according to a predefined trajectory following a registration process between the device's coordinate system and real-time CT images.
  Interventions: Device: XACT Robotic System

INTERVENTIONS:
Device: XACT Robotic System — CT-guided Minimally Invasive Procedures e.g., Biopsies

SUMMARY:
This is a prospective, single arm study, to evaluate the safety, effectiveness and usability of the XACT device. Subjects undergoing CT-guided, minimally invasive percutaneous lung procedures in the interventional radiology suite. eg. core, biopsy, will participate in the study. System and clinical accuracy will be the primary efficacy endpoint. Usability and safety will also be evaluated.

DETAILED DESCRIPTION:
This is a prospective, single-arm study is to evaluate the safety, effectiveness and usability of the XACT device. The study will be approved by the Institutional Review Board (IRB) at each of the participating centers prior to patient enrollment.

Subjects undergoing CT-guided, minimally invasive percutaneous lung procedures in the interventional radiology suite, e.g., core biopsy, fine needle aspiration (FNA), tumor ablation, etc., and willing to sign an informed consent document will be screened for compliance with the study inclusion and exclusion criteria.

A total of thirty (41) subjects will be enrolled in the study at 5 medical centers. The intention is to recruit subjects, which will cover a variety of CT-guided interventional lung procedures and a variety of different procedural tools that may be used with the device. Investigators will screen patients based on the inclusion/exclusion criteria described below and the subjects' demographic, general medical history, medical condition/indication, coagulation factors, concomitant medications and vital signs will be obtained.

The system accuracy will be the primary efficacy endpoint and is defined as the measured distance from the tip of the needle/tool to the target, once the XACT robot reaches the pre-defined target .

Clinical accuracy will be the secondary efficacy endpoint and is defined as the ability to place the instrument or procedural tool at a location suitable for the planned intervention. The investigator will review the final instrument position on the post-placement CT images to determine if the pre-operative planned target was reached. This information will be used to calculate success rate.

Additionally, the usability of the XACT device will be evaluated using a rating scale by assessing the ease of device setup, device operation, pre-operative planning, robot positioning, guiding and needle advancement. The total time of the procedure will be recorded, as will the number of CT scans performed and the radiation dose (DLP and CTDI).

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Subjects undergoing CT-guided, minimally invasive percutaneous procedures in the interventional radiology suite, e.g., core biopsy, fine needle aspiration (FNA), tumor ablation, etc.
* Subject is capable and willing to provide informed consent.
* Subject is capable and willing to adhere to the study procedures.

Exclusion Criteria:

* Subjects in whom the target is written 1 cm of a major blood vessel or major nerve.
* Subject with lesion in the central and peripheral nervous system and the spine.
* Subjects in whom the target is within 1 cm of a major blood vessel or major nerve.
* Subject with significant coagulopathy
* Subjects with a preexisting conditions, which, in the opinion of the investigator, may interfere with the conduct of the study.
* Subjects with an unstable medical condition, e.g. unstable hypertension, unstable cardiac disease, etc.
* Subjects who are uncooperative or cannot follow instructions.
* Subjects with a mental state that may preclude completion of the study procedure.
* Female subjects who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
System accuracy will be determined by the measured distance from the tip of the needle/tool to the target. | At the end of each interventional procedure, approximately 1 hour
  The primary endpoint of the study is to evaluate the system accuracy of the XACT System. System accuracy of the study will be determined by the measured distance from the tip of the needle/tool to the target, once the XACT Robot reaches the pre-defined target.

SECONDARY OUTCOMES:
Clinical accuracy of the study will be determined by the ability of the XACT system to reach the pre-defined target in each procedure. | At the end of each interventional procedure, approximately 1 hour
  The secondary endpoint of the study is to evaluate the clinical accuracy of the XACT system. Clinical accuracy of the study will be determined by the ability of the XACT system to reach the pre-defined target in each procedure.

OTHER OUTCOMES:
Device Usability | At the end of each interventional procedure, approximately 1 hour
  Usability of the XACT device performance in the hands of users will be evaluated using a rating scale for assessing the ease of device performance.
Evaluation of Safety | Through study completion (2 weeks)
  Evaluation of safety by assessing frequency, severity and causality of device related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ahava Stein, Study Director — A. Stein Regulatory Affairs Consulting Ltd.
Locations (2):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No